CLINICAL TRIAL: NCT05340140
Title: The Accuracy of Computer Aided Detection of Second Mesio-buccal Canal of Maxillary First Molars on CBCT Images Using Deep Learning Model (Artificial Intelligence): Diagnostic Accuracy Study
Brief Title: The Accuracy of Detection of Artificial Intelligence Second Mesio-buccal Canal of Maxillary First Molars on CBCT Images
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Arwa Mousa, lecturer of oral and maxillofacial radiology, faculty of dentistry, Cairo University
Other Study IDs: CBCT AI 7-1-1
Record Dates: First submitted 2022-04-15; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Artificial Intelligence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CBCT Images of Maxillary 1st molars
  Interventions: Diagnostic Test: deep learning model

INTERVENTIONS:
Diagnostic Test: deep learning model — deep learning model developed by computer science expert and based on convolution neural network , and trained by our datasets.
  Other Names: artificial intelligence tool

SUMMARY:
CAD systems are computer applications that assist in the detection and/or diagnosis of diseases by providing an unbiased "second opinion" to the image interpreter, aiming at improving accuracy and reducing time for analysis. With the rapid growth of Deep Learning (DL) algorithms in image-based applications, CAD systems can now be trained by DL to provide more advanced capability (ie, the capability of artificial intelligence [AI]) to best assist clinicians.

DETAILED DESCRIPTION:
Countless studies and discussions have been based on the existence of a second canal in the mesiobuccal (MB) root of the maxillary molars , since it is strongly believed that one of the foremost reasons for endodontic failure in maxillary first molars is the difficulty of detecting and treating those second mesiobuccal (MB2) canals .The literature reveals that although MB2 canals of maxillary first molars have been found in more than 70% of in vitro studies , they were detected clinically in less than 40% of cases . Cone beam computed tomography (CBCT) is an imaging modality in the field of endodontics that has several advantages, including the ability to perform three-dimensional (3D) imaging of root canal systems with lower radiation doses, higher resolution, and no superimposition . Researchers have evaluated the efficiency of CBCT when it comes to identifying MB2 canals, and CBCT has been suggested to be a reliable method for the detection of these canals. However, in clinically relevant situations, such a smaller lesions on root-filled teeth, CBCT accuracy is greatly reduced (sensitivity 0.63, specificity 0.69) . Moreover, clinician dependent interpretation of CBCT imaging still suffers from low inter- and intra-observer agreement.

Computer-aided detection and diagnosis (CAD) has been widely applied to biomedical image analysis outside of dentistry .

ELIGIBILITY:
Inclusion Criteria:

* • CBCT scans showing erupted maxillary 1st molar.

  * Vovel size not exceeding 0.1mm.
  * Maxillary molars showing complete root formation.
  * Carious or Non-carious tooth.

Exclusion Criteria:

* • Maxillary first molars with developmental anomalies, external or internal root resorption, root canal calcification, previous root canal treatment, post restorations, and/or root caries.

  * CBCT images of sub-optimal quality or artifacts / high scatter interfering with proper assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CBCT scans showing maxillary first molars with resolution not more than 0.1 mm voxel size.The CBCT data of this study will be obtained from the CBCT data base available at the department of Oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University, Cairo, Egypt and from multiple private radiology centres using the same machine brand with the same parameters. CBCT scans of Egyptian patients who have already been subjected to CBCT examination as part of their dental diagnosis and/or treatment planning from January 2020 to December 2022 will be included according to the proposed eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
accuracy of detection of MB2 | baseline
  detection of MB2 on CBCT images of maxillary first molars using deep learning model

CONTACTS AND LOCATIONS:
Overall Officials: Enas Anter, Ph.D, Study Director — Cairo University
Locations (1):
- Faculty of dentistry cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Blattner TC, George N, Lee CC, Kumar V, Yelton CD. Efficacy of cone-beam computed tomography as a modality to accurately identify the presence of second mesiobuccal canals in maxillary first and second molars: a pilot study. J Endod. 2010 May;36(5):867-70. doi: 10.1016/j.joen.2009.12.023. Epub 2010 Feb 21. PMID 20416435
- [Background] Kulild JC, Peters DD. Incidence and configuration of canal systems in the mesiobuccal root of maxillary first and second molars. J Endod. 1990 Jul;16(7):311-7. doi: 10.1016/s0099-2399(06)81940-0. PMID 2081944
- [Background] Alacam T, Tinaz AC, Genc O, Kayaoglu G. Second mesiobuccal canal detection in maxillary first molars using microscopy and ultrasonics. Aust Endod J. 2008 Dec;34(3):106-9. doi: 10.1111/j.1747-4477.2007.00090.x. PMID 19032644
- [Background] Gorduysus MO, Gorduysus M, Friedman S. Operating microscope improves negotiation of second mesiobuccal canals in maxillary molars. J Endod. 2001 Nov;27(11):683-6. doi: 10.1097/00004770-200111000-00008. PMID 11716081
- [Background] Weine FS, Hayami S, Hata G, Toda T. Canal configuration of the mesiobuccal root of the maxillary first molar of a Japanese sub-population. Int Endod J. 1999 Mar;32(2):79-87. doi: 10.1046/j.1365-2591.1999.00186.x. PMID 10371900
- [Background] Ekert T, Krois J, Meinhold L, Elhennawy K, Emara R, Golla T, Schwendicke F. Deep Learning for the Radiographic Detection of Apical Lesions. J Endod. 2019 Jul;45(7):917-922.e5. doi: 10.1016/j.joen.2019.03.016. Epub 2019 Jun 1. PMID 31160078
- [Background] Hiraiwa T, Ariji Y, Fukuda M, Kise Y, Nakata K, Katsumata A, Fujita H, Ariji E. A deep-learning artificial intelligence system for assessment of root morphology of the mandibular first molar on panoramic radiography. Dentomaxillofac Radiol. 2019 Mar;48(3):20180218. doi: 10.1259/dmfr.20180218. Epub 2018 Nov 9. PMID 30379570
- [Background] Orhan K, Bayrakdar IS, Ezhov M, Kravtsov A, Ozyurek T. Evaluation of artificial intelligence for detecting periapical pathosis on cone-beam computed tomography scans. Int Endod J. 2020 May;53(5):680-689. doi: 10.1111/iej.13265. Epub 2020 Feb 3. PMID 31922612
- [Derived] Mansour S, Anter E, Mohamed AK, Dahaba MM, Mousa A. Two step approach for detecting and segmenting the second mesiobuccal canal of maxillary first molars on cone beam computed tomography (CBCT) images via artificial intelligence. BMC Oral Health. 2025 Sep 8;25(1):1404. doi: 10.1186/s12903-025-06796-4. PMID 40926256